CLINICAL TRIAL: NCT00395577
Title: A Phase 2, 12-Week, Randomized, Placebo-Controlled Study to Evaluate the Antiinflammatory Effects of VX-702 When Administered Concomitantly With Methotrexate
Brief Title: A Study in Rheumatoid Arthritis With an Investigational Oral p38 MAP Kinase Inhibitor VX-702
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX06-702-304
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — VX 702

INTERVENTIONS:
Drug: VX-702

SUMMARY:
The purpose of this study is to assess the safety and effects of VX-702 in subjects with moderate to severe rheumatoid arthritis and who are taking the drug methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 to 75 years of age with active RA
* Must have been taking MTX for at least 6 months
* No concurrent DMARD treatment (other than a stable dose of MTX)

Exclusion Criteria:

* Planned major surgery (e.g., joint replacement) within the duration of the treatment period of the study
* Treated with intra-articular injections of corticosteroids within 28 days prior to Day 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of VX-702 administered with concomitant methotrexate (MTX), and MTX alone

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of VX-702 administered with concomitant MTX, and MTX alone

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kauffman, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (17):
- Bulgaria (4):
  - Call For Information, Dimitrovgrad
  - Call For Information, Pleven
  - Call For Information, Sofia
  - Call For Information, Veliko Tarnovo
- Croatia (2):
  - Call For Information, Osijek
  - Call For Information, Zagreb
- Poland (4):
  - Call For Information, Bytom
  - Call For Information, Krakow
  - Call for Information, Torun
  - Call For Information, Żyrardów
- Russia (3):
  - Call For Information, Novosibirsk
  - Call For Information, Saint Petersburg
  - Call For Information, Saratov
- Serbia and Montenegro (3):
  - Call For Information, Belgrade
  - Call For Information, Niska Banja
  - Call For Information, Zemun
- Call For Information, Ljubljana, Slovenia

REFERENCES:
- [Derived] Damjanov N, Kauffman RS, Spencer-Green GT. Efficacy, pharmacodynamics, and safety of VX-702, a novel p38 MAPK inhibitor, in rheumatoid arthritis: results of two randomized, double-blind, placebo-controlled clinical studies. Arthritis Rheum. 2009 May;60(5):1232-41. doi: 10.1002/art.24485. PMID 19404957